CLINICAL TRIAL: NCT06910670
Title: Implementing a Randomized Control Trial to Test the Expanded Web-based Decision Aid
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 202409214; U2CCA252981 (NIH)
Record Dates: First submitted 2025-03-20; First posted 2025-04-04 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Cholangiocarcinoma; Colorectal Cancer; Multiple Myeloma
Keywords: Genetic testing; Decision aid; Participant engagement
MeSH Terms: conditions — Cholangiocarcinoma; Colorectal Neoplasms; Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention: Genetics Advisor Online Tool (Experimental): The Intervention group will receive the expanded Genetics Advisor decision aid.
  Interventions: Other: Genetics Advisor Decision Aid
- Control: Standard developed materials (Active Comparator): The control group will receive a description of each type of genomic sequencing result they could receive using the standard informed consent process for the return-of-results protocol.

INTERVENTIONS:
Other: Standard developed materials — Participants will be given the option to receive different types of results from genomic sequencing. The choices available to them will be explained by research staff following a script that describes what each type of result means. Participants will be able to choose to receive: (1) no results, or any combination of (2) biomarker information from cancer cells, (3) inherited mutations related to cancer, and (4) inherited mutations related to other medical issues. These choices will be presented to them via a discussion with study staff with accompanying paper information
Other: Genetics Advisor Decision Aid — Participants will be given the option to receive different types of results from genomic sequencing. The participants will be given access to a web-based decision aid that elicits participants' values and preferences for receiving results from cancer genomic sequencing to guide them making a decision about what types of results they would like to receive. Participants will be able to choose to receive: (1) no results, or any combination of (2) biomarker information from cancer cells, (3) inherited mutations related to cancer, and (4) inherited mutations related to other medical issues.
  Arms: Intervention: Genetics Advisor Online Tool

SUMMARY:
The overall goal of the randomized control trial (RCT) will be to evaluate the efficacy of modifications to a web-based tool for patient decision-making regarding return of genomic results that will more closely focus on rare cancers. Participants will be given access to a web-based decision aid (or a standard control) that guides participants in making decisions about what type of genomic results they would like to receive from testing performed in the PE-CGS study (NCT06340646).

ELIGIBILITY:
Eligibility Criteria:

* Enrolled in the WU-PE-CGS study (IRB#202106129); that eligibility entails:

  * Diagnosis of cholangiocarcinoma
  * Diagnosis of multiple myeloma, must be African American
  * Diagnosis of colorectal cancer, must be African American and age 65 or older at time of diagnosis
* At least 18 years old.
* Able to understand an IRB-approved informed consent document and agree to participation
* Have access to a personal computer, tablet or mobile device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in self-efficacy about genomic test results | Baseline, after viewing assigned materials (day 1), and 3-months after enrollment
  7-item, Likert scale. This scale has 5 points ranging from strongly disagree to strongly agree. 1= Strongly disagree, 2= Disagree, 3= Neither Agree nor Disagree, 4= Agree, 5= Strongly Agree. All items are scored such that 'strongly agree' reflects a correct response and 'agree' reflects a less confident correct response in the correct direction. This will be scored by adding up the numbers for each of the 7 items regarding self-efficacy. The total score ranges from 7 to 35. A higher score for the participant represents higher participant self-efficacy.

SECONDARY OUTCOMES:
Change in decisional conflict | After viewing assigned materials (day 1) and 3-months after enrollment
  17-item, Likert scale. This scale has 5 points ranging from strongly agree to strongly disagree. 1=Strongly Agree, 2=Agree, 3=Neither Agree nor Disagree, 4=Disagree, 5=Strongly Disagree. All items are scored such that 'strongly disagree' reflects an incorrect response and 'disagree' reflects a less confident incorrect response in the incorrect direction. This will be scored by adding up the numbers for each of the 17 items regarding decisional conflict. The total score ranges from 17 to 85. The higher score for the participant represents higher participant decisional conflict.
Change in knowledge of clinical genetic testing | After viewing assigned materials (day 1) and 3-months after enrollment
  12-item, Likert scale. This scale has 5 points ranging from strongly agree to strongly disagree. 1=Strongly Agree, 2=Agree, 3=Neither Agree nor Disagree, 4=Disagree, 5=Strongly Disagree for items (4, 6-12) are scored such that 'strong disagree' reflects a correct response and 'somewhat disagree' reflects a less confident correct response in the correct direction. Negatively worded items (items 1, 2, 3, 5) are reverse scored so that "strongly agree' reflected a correct response and 'somewhat agree' reflected a less confident response in the correct direction. This will be scored by adding up the numbers for each of the 11 items regarding participant knowledge of clinical genetic testing. The total score ranges from 12 to 60. A higher score for the participant represents higher participant knowledge.
Change in expectations for potential benefits of cancer genomic sequencing | After viewing assigned materials (day 1) and 3-months after enrollment
  Participants will rate their expectation for 6 potential benefits of cancer genomic sequencing on a 4-point scale ranging from extremely unlikely to extremely likely. . 1= Extremely unlikely, 2= Unlikely, 3= Likely, 4= Extremely likely. This will be scored by adding up the numbers for each of the 6 items regarding participant expectations of benefit. The total score ranges from 6 to 24. A higher score for the participant represents higher levels of expectations.
Decisional conflict scores categorized by demographic factors | After viewing assigned materials (day 1) and 3-months after enrollment
  17-item, Likert scale. This scale has 5 points ranging from strongly agree to strongly disagree. 1=Strongly Agree, 2=Agree, 3=Neither Agree nor Disagree, 4=Disagree, 5=Strongly Disagree. All items are scored such that 'strongly disagree' reflects an incorrect response and 'disagree' reflects a less confident incorrect response in the incorrect direction. This will be scored by adding up the numbers for each of the 17 items regarding decisional conflict. The total score ranges from 17 to 85. The higher score for the participant represents higher participant decisional conflict.
  Demographic factors include age, race, SES, and geographic residence.
Knowledge scores categorized by demographic factors | After viewing assigned materials (day 1) and 3-months after enrollment
  12-item, Likert scale. This scale has 5 points ranging from strongly agree to strongly disagree. 1=Strongly Agree, 2=Agree, 3=Neither Agree nor Disagree, 4=Disagree, 5=Strongly Disagree for items (4, 6-12) are scored such that 'strong disagree' reflects a correct response and 'somewhat disagree' reflects a less confident correct response in the correct direction. Negatively worded items (items 1, 2, 3, 5) are reverse scored so that "strongly agree' reflected a correct response and 'somewhat agree' reflected a less confident response in the correct direction. This will be scored by adding up the numbers for each of the 11 items regarding participant knowledge of clinical genetic testing. The total score ranges from 12 to 60. A higher score for the participant represents higher participant knowledge.
  Demographic factors include age, race, SES, and geographic residence.
Decisional conflict scores categorized by genomic literacy | After viewing assigned materials (day 1) and 3-months after enrollment
  Genomic literacy will be measured at baseline. 14 items. For 7 items participants will rate their familiarity with genetic terminology on a 7 point scale ranging from strongly disagree to strongly agree. 1= Strongly disagree, 7= Strongly agree. This portion ill be scored by adding up the numbers for each of these 7 items. The total score on this portion ranges from 7 to 49. An additional 7 questions ask participants to fill in a missing word in a statement about genetics. These 7 items are multiple-choice questions and are scored by adding up the number of correct answers. The score on this portion ranges from 0 to 7.
Knowledge scores categorized by genomic literacy | After viewing assigned materials (day 1) and 3-months after enrollment
  Genomic literacy will be measured at baseline. 14 items. For 7 items participants will rate their familiarity with genetic terminology on a 7 point scale ranging from strongly disagree to strongly agree. 1= Strongly disagree, 7= Strongly agree. This portion ill be scored by adding up the numbers for each of these 7 items. The total score on this portion ranges from 7 to 49. An additional 7 questions ask participants to fill in a missing word in a statement about genetics. These 7 items are multiple-choice questions and are scored by adding up the number of correct answers. The score on this portion ranges from 0 to 7.
Decisional conflict scores categorized by genomic sequencing testing attitudes | After viewing assigned materials (day 1) and 3-months after enrollment
  Genomic sequencing testing attitudes is measured at baseline. 6-items. This scale has 4 points ranging from 'strongly disagree' to 'strongly agree'. 1= Strongly disagree, 4=Strongly agree. This is scored by adding up the numbers for each of the 6 items. The score ranges from 6 to 24. A higher score indicates a higher participant level of trust in genomic research participation.
Knowledge scores categorized by genomic sequencing testing attitudes | After viewing assigned materials (day 1) and 3-months after enrollment
  Genomic sequencing testing attitudes is measured at baseline. 6-items. This scale has 4 points ranging from 'strongly disagree' to 'strongly agree'. 1= Strongly disagree, 4=Strongly agree. This is scored by adding up the numbers for each of the 6 items. The score ranges from 6 to 24. A higher score indicates a higher participant level of trust in genomic research participation.
Decisional conflict scores categorized by clinical characteristics | After viewing assigned materials (day 1) and 3-months after enrollment
  7-item, Likert scale. This scale has 5 points ranging from strongly disagree to strongly agree. 1= Strongly disagree, 2= Disagree, 3= Neither Agree nor Disagree, 4= Agree, 5= Strongly Agree. All items are scored such that 'strongly agree' reflects a correct response and 'agree' reflects a less confident correct response in the correct direction. This will be scored by adding up the numbers for each of the 7 items regarding self-efficacy. The total score ranges from 7 to 35. A higher score for the participant represents higher participant self-efficacy.
  Clinical characteristics include cancer type, stage at diagnosis, and primary treatment.
Knowledge scores categorized by clinical characteristics | After viewing assigned materials (day 1) and 3-months after enrollment
  12-item, Likert scale. This scale has 5 points ranging from strongly agree to strongly disagree. 1=Strongly Agree, 2=Agree, 3=Neither Agree nor Disagree, 4=Disagree, 5=Strongly Disagree for items (4, 6-12) are scored such that 'strong disagree' reflects a correct response and 'somewhat disagree' reflects a less confident correct response in the correct direction. Negatively worded items (items 1, 2, 3, 5) are reverse scored so that "strongly agree' reflected a correct response and 'somewhat agree' reflected a less confident response in the correct direction. This will be scored by adding up the numbers for each of the 11 items regarding participant knowledge of clinical genetic testing. The total score ranges from 12 to 60. A higher score for the participant represents higher participant knowledge.
  Clinical characteristics include cancer type, stage at diagnosis, and primary treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Erin Linnenbringer, Ph.D., MS, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
Will share all data, software and know-how generated during the course of this work, without limitations except as prevented by prior agreement. This will include both the final datasets, as well as the data necessary to complete the aims. Will disseminate results from this research through presentations at public lectures, scientific institutions and meetings, and/or publication in major journals. All final peer-reviewed manuscripts that arise from this proposal will be submitted to the digital archive PubMed Central. Wherever applicable, data will be deposited to appropriate public repositories.
  All participants whose genomic data are collected will be consented for broad data sharing, and their genomic data will be included in the study deposits. Data documentation and de-identified data will be deposited for sharing along with phenotypic data, which includes demographics and diagnosis, consistent with applicable laws and regulations.
Supporting Information: Study Protocol, SAP
Time Frame: The investigators agree to deposit data into database of Genotypes and Phenotypes (dbGaP) repository after data cleaning and quality control as soon as possible but no later than within three months, or upon acceptance of the data for publication, or public disclosure of a submitted patent application, whichever is earlier. When data are released from dbGaP, the data will be made available to the Genomic Data Commons (GDC).
Access Criteria: The investigators agree that they will identify where the data will be available (dbGaP and GDC) and how to access the data in any publications and presentations that they author or co-author about these data, as well as acknowledge the repository and funding source in any publications and presentations. As they will be using the database of Genotypes and Phenotypes (dbGaP), which is an NIH-funded repository, this repository has policies and procedures in place that will provide data access to qualified researchers, fully consistent with NIH data sharing policies and applicable laws and regulations.

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu